CLINICAL TRIAL: NCT02336945
Title: Glucose Variability Pilot Study for the Abbott Sensor Based Glucose Monitoring System-Professional
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-RES-14137
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 diabetes: Subjects with type 2 diabetes who meet one of the therapy conditions
  Interventions: Device: Abbott Sensor Based Glucose Monitoring System-Professional

INTERVENTIONS:
Device: Abbott Sensor Based Glucose Monitoring System-Professional — Subjects will wear 2 glucose sensors while going about daily activities and adhering to establish diabetes treatment plan. This is not a treatment study.
  Other Names: FreeStyle Libre Pro

SUMMARY:
This is a multi-center, prospective, non-pivotal, single arm, non-significant risk evaluation the Abbott Sensor Based Glucose Monitoring System - Pro across different stages of T2 diabetes management. This is a non-significant risk study.

DETAILED DESCRIPTION:
Subjects will wear two Sensors, one applied to the back of each upper arm, for a period of 14 days. Subjects will wear the Sensor while going about their normal daily activities during the home use period. Subjects will not be able to see any glucose data. The devices will be removed at the completion of the final study visit.

Data obtained from the Reader and reports generated by the system will not be used by the subject or the research team members to determine treatment. Subjects must adhere to their diabetes clinical management plan established prior to the study.

No additional medical care will be provided to study subjects following study completion other than care related to the follow up and treatment of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must have diagnosis of type 2 diabetes prior to enrollment.
3. Subject must have been on current treatment regimen for at least 6 months prior to enrollment and must remain on therapy regimen for the duration of the study (subjects diagnosed within last 6 months must be on no medication both prior to and throughout the study to enroll).
4. HbA1c greater than or equal to 6.0% or less than or equal to 12.0% as demonstrated by lab HbA1c result obtained within the last 6 months.

   1. Subjects with HbA1c <7.5% will be excluded from the study if the subject's intended therapy group for enrollment requires an HbA1c ≥7.5%.
   2. For therapy groups enrolling 12 subjects with HbA1c of <7.5% and 12 subjects with HbA1c of ≥7.5%, subjects with an HbA1c level within each respective range will be excluded from the study once the enrollment goal of that HbA1c range has been met.
   3. If no HbA1c taken within the last six months is available, a new laboratory HbA1c value must be obtained prior to Sensor application.
5. Subject must be able to read and understand English.
6. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol
7. In the investigators opinion, the subject must be compliant with their diabetes management plan and must be able to adhere to medication regimen throughout study.
8. Subject must be available to participate in all study visits.
9. Subject must be willing and able to provide written signed and dated informed consent.

Exclusion Criteria:

1. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
2. Subject is pregnant, is attempting to conceive or is not willing and able to practice birth control during the study duration (applicable to female subjects only).
3. Subject has skin lesions, scarring, redness, infection or edema at the application sites that could interfere with device placement or the accuracy of interstitial glucose measurements.
4. Subject currently is participating in another clinical trial.
5. Subject has X-ray, MRI or CT appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
6. HbA1c of less than 6.0% or greater than 12.0% as demonstrated by lab HbA1c result obtained within the last 6 months.
7. Enrollment goal of Subject's intended therapy group has been met.
8. Subject is unsuitable for participation due to any other cause as determined by the Investigator.
9. Subject is currently on one of the following treatments or treatment combinations:

   1. Metformin + Sulfonylurea + DPP-4 Inhibitor
   2. Sulfonylurea + DPP-4 Inhibitor
   3. Metformin + Sulfonylurea + GLP-1 Receptor Agonist
   4. Sulfonylurea + GLP-1 Receptor Agonist
   5. Metformin + Sulfonylurea + SGLT-2
   6. Sulfonylurea + SGLT-2
   7. Metformin + SGLT-2 + Insulin
   8. SGLT-2 + Insulin
   9. NPH Insulin (with exception of NPH insulin present in premix formulations)
   10. Rapid acting insulin (with exception of rapid acting insulin present in premix formulations)
   11. Four (4) or more diabetes therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 2 diabetes who meet one of the therapy groups
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Glucose variability as measured by AGP Interquartile Range, (IQR) obtained via System-Pro Sensor. | 2 weeks

SECONDARY OUTCOMES:
Assessment of ambulatory glucose profiles (AGPs) generated by the Software | 2 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Unger Primary Care Medical Center & Catalina Research Institute, Chino, California
  - Dr. Deanna Cheung, Long Beach, California
  - University of California San Diego Veterns Affairs Medical Center, San Diego, California
  - Henry Ford Medical Center, Detroit, Michigan
  - St. Luke's Endocrinology and Diabetes, Kansas City, Missouri
  - Duke Southern Regional AHEC, Fayetteville, North Carolina
  - Diabetes America- Pearland, Pearland, Texas